CLINICAL TRIAL: NCT02108886
Title: Pilot Study Testing a New Strategy for Management of Spontaneous Preterm Birth.
Acronym: EAU2-Mtlk
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, MD, PhD, Dr, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-143
Record Dates: First submitted 2013-01-15; First posted 2014-04-09 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Preterm Labor
Keywords: preterm labor; montelukast; uterine contractions
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — montelukast; Urination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Experimental): Intervention group
  Interventions: Drug: Montelukast; Other: urine and vaginal secretions sampling
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Other: urine and vaginal secretions sampling

INTERVENTIONS:
Drug: Montelukast — 10 mg of Montelukast per day, from admission for preterm labor until delivery or 35 weeks of pregnancy.
  Other Names: Singulair
  Arms: Montelukast
Drug: Placebo — empty capsule filled with sugar
  Arms: Placebo
Other: urine and vaginal secretions sampling — Urine and vaginal secretions sampling, once a week in both groups

SUMMARY:
Preterm birth is a major public health problem, and actual treatments are not very efficient. The purpose of this study is to test the efficiency of a combined use of Montelukast and Nifedipine to treat preterm labor. Investigators aim to reduce uterine contractions more efficiently than with the use of Nifedipine only.

DETAILED DESCRIPTION:
An inflammatory process is involved in 60% of preterm births. Moreover, investigators previously demonstrated that enzymes of lipoxygenase pathway are present in uterine smooth muscle, and that an additive tocolytic effect can be obtained from the combined use of Montelukast and Nifedipine.

Methods:

This is a double-blinded randomized controlled assay performed at the CHUS on two groups of 50 women. Women will be selected when admitted for preterm labor with a gestational age between 26 and 34 weeks.

The first group will receive Nifedipine for 48 hours, as described by the standard protocol at the CHUS, in addition to 10 mg of Montelukast per day, until delivery or 35 weeks of pregnancy.

The second group will receive Nifedipine for 48 hours, as described by the standard protocol at the CHUS, in addition to a placebo per day, until delivery or 35 weeks of pregnancy.

Cervical secretions and urine will be sample at the admission, after one week and every two weeks during treatment.

ELIGIBILITY:
Inclusion Criteria:

* women with 24-34 weeks of pregnancy
* indication for tocolysis

Exclusion Criteria:

* preterm labor before 26 or after 34 weeks of pregnancy
* minor patients
* patients with other obstetrical pathology
* twin pregnancies
* fetal distress
* severe congenital fetal malformation
* anti-phospholipid syndrome
* lupus
* gestational diabetes
* nephropathy
* congenital heart disease
* obvious causes of infection associated with prematurity
* patients with viral infections (HIV, hepatitis)
* patients already treated with Montelukast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Time between beginning of treatment and delivery | until delivery (max 17 weeks)

SECONDARY OUTCOMES:
preterm birth | until delivery (max 13 weeks)
  birth before 37 weeks of gestation
chorio decidual infection | between inclusion and delivery (max 17 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada